CLINICAL TRIAL: NCT04891978
Title: Implementation of the US PRECISION AIRQ, Asthma Checklist, and Educational Resources (PRECISION Program) Into Clinical Practice Using Telehealth and In-Person Platforms
Brief Title: US PRECISION Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D2287L00028
Record Dates: First submitted 2021-03-29; First posted 2021-05-19 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AIRQ, Asthma Checklist, and PRECISION Program (Experimental): All participants in the trial will be given the behavioral interventions which include the AIRQ tool, the Asthma Checklist tool, and the PRECISION program educational resources.
  Interventions: Behavioral: AIRQ; Behavioral: Asthma Checklist; Behavioral: PRECISION Program (Educational Resources)

INTERVENTIONS:
Behavioral: AIRQ — A validated tool designed to identify patients who may be at risk for adverse outcomes from uncontrolled asthma.
Behavioral: Asthma Checklist — A validated, 3-page tool, based on GINA and NAEPP guidelines to assist providers with recognition, evaluation, and optimization of all patients with asthma. In this study, healthcare providers will be required to complete the assess component (page 1) of the Asthma Checklist .
Behavioral: PRECISION Program (Educational Resources) — Educational resources accessible to all providers in the study. There are provider-facing and patient-facing educational materials that can be accessed during the patient visit or as resources for before/after visits. Resources can be downloaded and sent to patients per the discretion of providers.

SUMMARY:
The primary objective of this community program intervention study is to assess the process and potential benefits of integrating the AIRQ®, Asthma Checklist, and educational resources (PRECISION program) into clinical practice using either in-person or telehealth visits.

The secondary objectives are to assess asthma patients' clinic visit experiences when the AIRQ, the Asthma Checklist, and educational resources (PRECISION program) are utilized as part of a telehealth or in-person visit with their HCP, and to explore change in AIRQ scores from the initial visit to follow-up visit(s) (when available).

DETAILED DESCRIPTION:
This community program intervention study will examine the process of integrating the AIRQ, Asthma Checklist, and educational resources (PRECISION program) into clinical practice using either in-person or telehealth visits. Providers use of patients' responses to the AIRQ, Asthma Checklist, and educational resources to guide treatment and asthma work-up and management also will be examined. The study duration is 12-months, with study enrollment lasting nine (9) months for each site (implementation stage), and an additional three (3) months of follow-up to assess the sustainability of using the PRECISION program in clinical practice (sustainability stage). The nine-month implementation stage will allow for the recruitment of approximately 50 patients at each site (maximum of 75 patients at each site) for an initial study visit, plus the potential for follow-up visit(s). The three-month sustainability stage will allow for sites to continue to implement the PRECISION program in their clinical practice and for sites to describe any continued benefits of using the PRECISION program at their site.

Approximately fifteen (15) to twenty (20) clinical sites will be recruited to participate in this study, categorized into the following four practice clusters: (1) primary care site (e.g., private practice, FQHC; (2) specialty care site (pulmonary, asthma/immunology); and (3) novel sites (e.g., pharmacy, nurse practitioners, nurse educators, prescribers and Non-prescribers, telehealth component of Allergy and Asthma Network. While all sites will be able to conduct both in-person and telehealth visits, sites will aim to conduct a minimum of approximately 25% of their initial patient visit using a telehealth platform. Both platforms (in-person and telehealth) can be used for the follow-up visit(s) for all practice types.

ELIGIBILITY:
Inclusion Criteria:

* >= 13 years of age at the time of enrollment
* Diagnosis of HCP-confirmed asthma
* Able to read, understand and speak English or Spanish sufficiently self-complete or be administered the AIRQ via telephone, desktop, or mobile device (e.g., smartphone, iPad)
* Provide consent (adults/parents/guardians) and assent (age 13-17 years) to participate in the study.

Exclusion Criteria:

* Current diagnosis of active COPD or any lower respiratory diagnosis other than asthma
* Has a cognitive impairment, hearing difficulty, acute psychopathology, medical condition, or insufficient knowledge of the English or Spanish language that, in the opinion of the investigator, would interfere with his or her ability to agree to participate and/or complete the AIRQ or other study questionnaires

Ages: 13 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 857 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Research Site, Birmingham, Alabama
  - Research Site, Leesburg, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Fort Wayne, Indiana
  - Research Site, Tewksbury, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Cornwall-on-Hudson, New York
  - Research Site, Rochester, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, San Antonio, Texas
  - Research Site, Vienna, Virginia
  - Research Site, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Murphy KR, Chipps B, Beuther DA, Wise RA, McCann W, Gilbert I, Eudicone JM, Gandhi HN, Harding G, Coyne KS, Zeiger RS; US PRECISION Advisory Board. Development of the Asthma Impairment and Risk Questionnaire (AIRQ): A Composite Control Measure. J Allergy Clin Immunol Pract. 2020 Jul-Aug;8(7):2263-2274.e5. doi: 10.1016/j.jaip.2020.02.042. Epub 2020 May 6. PMID 32387166
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287L00028&attachmentIdentifier=ca020a9f-15e9-4d3f-87a6-45c3be534fb5&fileName=D2287L00028_Implementation_Study_Report_Synopsis_Final_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen sites in the US were selected (6 primary care, 6 specialty care, 1 novel site) to implement the PRECISION program. Clinic staff invited patients ≥13 years old with HCP-confirmed asthma diagnosis who were presenting for a telehealth or in-person visit to complete the AIRQ. Each primary and specialty site aimed to recruit approximately 50 patients, up to 100 maximum. The novel site aimed to recruit 150 patients. Patients were recruited between April 2021 and February 2022.
Units Other Than Participants: Sites
Groups:
- Primary Care Sites: e.g., private practice, FQHC
- Specialty Care Sites: e.g., pulmonary, asthma/immunology
- Novel Site: e.g., telehealth component of Allergy and Asthma Network
Period: Baseline
Arm/Group | Primary Care Sites | Specialty Care Sites | Novel Site
Started (Number of patients who consented to take part) | 434; 6 Sites | 281; 6 Sites | 142; 1 Sites
Completed (Number of patients who were enrolled in the study (consented, completed baseline visit and completed baseline AIRQ)) | 431; 6 Sites | 280; 6 Sites | 133; 1 Sites
Not Completed | 3; 0 Sites | 1; 0 Sites | 9; 0 Sites
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Missing AIRQ | 1 | 0 | 0
Not completed — Did not attend a baseline visit | 0 | 0 | 9
Period: Follow-up
Arm/Group | Primary Care Sites | Specialty Care Sites | Novel Site
Started (Patients who completed the initial visit) | 431; 6 Sites | 280; 6 Sites | 133; 1 Sites
Completed (Patients who completed a follow-up visit) | 145; 4 Sites | 100; 5 Sites | 126; 1 Sites
Not Completed | 286; 2 Sites | 180; 1 Sites | 7; 0 Sites

BASELINE CHARACTERISTICS:
Population: Baseline patient population from primary care, specialty care and novel sites who completed the AIRQ
Units Other Than Participants: Sites
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Sites | Specialty Care Sites | Novel Site | Total
Number analyzed (Participants) | 431 | 280 | 133 | 844
Number analyzed (Sites) | 6 | 6 | 1 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (18.8) | 46.9 (19.0) | 38.9 (14.2) | 45.4 (18.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 296 | 202 | 95 | 593
  Male | 134 | 77 | 38 | 249
  Other/non-binary | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 14 | 1 | 106
  Not Hispanic or Latino | 302 | 251 | 8 | 561
  Unknown or Not Reported | 38 | 15 | 124 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 57 | 4 | 0 | 61
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 0 | 4
  Black or African American | 75 | 42 | 2 | 119
  White | 254 | 217 | 7 | 478
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 40 | 15 | 124 | 179
Clinician's rating of patient's asthma severity [Count of Participants; unit: Participants]
  Intermittent | 206 | 30 | 42 | 278
  Mild persistent | 100 | 61 | 23 | 184
  Moderate persistent | 112 | 117 | 43 | 272
  Severe persistent | 13 | 71 | 25 | 109
  Missing | 0 | 1 | 0 | 1
AIRQ Control Categories [Count of Participants; unit: Participants]
  Well controlled (0-1) | 214 | 121 | 23 | 358
  Not well controlled (2-4) | 144 | 80 | 41 | 265
  Very poorly controlled (5-10) | 73 | 79 | 69 | 221

OUTCOME MEASURES:

1. Primary Outcome: Percentage Endorsement of Responses by Site HCPs for Each Categorical Item on the Post-study Survey Relating to Overall Ease of Implementing AIRQ Into Clinical Practice.
Description: The post-study HCP survey includes questions regarding the implementation of the PRECISION program (e.g., how would you rate the overall ease of implementing the AIRQ into your clinical practice using the telehealth platform?)
Time Frame: Post-study survey was completed between 5 weeks and 50.6 weeks of last patient end of follow-up across sites; end of follow up was 36 weeks from last patient enrolled at site (or 6 weeks for the novel care site).
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Groups:
- Novelty Care Site: e.g., telehealth component of Allergy and Asthma Network
- Total: All sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Sites
  Overall ease of implementing AIRQ into clinical practice using telehealth platform: Very easy | 1 | 3 | 1 | 5
  Overall ease of implementing AIRQ into clinical practice using telehealth platform: Somewhat easy | 4 | 2 | 0 | 6
  Overall ease of implementing AIRQ into clinical practice using telehealth platform: Difficult | 0 | 1 | 0 | 1
  Overall ease of implementing AIRQ into clinical practice using telehealth platform: Very Difficult | 0 | 0 | 0 | 0
  Overall ease of implementing AIRQ into clinical practice using telehealth platform: Missing | 1 | 0 | 0 | 1
  Overall ease of implementing AIRQ into clinical practice during an in-person visit: Very easy | 3 | 5 | 0 | 8
  Overall ease of implementing AIRQ into clinical practice during an in-person visit: Somewhat easy | 3 | 1 | 0 | 4
  Overall ease of implementing AIRQ into clinical practice during an in-person visit: Difficult | 0 | 0 | 0 | 0
  Overall ease of implementing AIRQ into clinical practice during an in-person visit: Very Difficult | 0 | 0 | 0 | 0
  Overall ease of implementing AIRQ into clinical practice during an in-person visit: Missing | 0 | 0 | 1 | 1

2. Primary Outcome: Percentage Endorsement of Responses by Site HCPs for the Categorical Item on the Post-study Survey Relating to How Much the AIRQ Helped Manage Patients
Description: The post-study HCP survey includes questions regarding the implementation of the PRECISION program at the site (e.g., Did AIRQ help you manage your patients?)
Time Frame: as for outcome 1
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Sites
  Yes very much | 5 | 0 | 0 | 5
  Yes somewhat | 1 | 5 | 1 | 7
  Not at all | 0 | 1 | 0 | 1

3. Primary Outcome: Percentage Endorsement of Responses by Site HCPs for the Categorical Item on the Post-study Survey Relating to Whether the AIRQ Helped Identify Patients at Risk for Adverse Asthma Health Outcomes
Description: The post-study HCP survey includes questions regarding the implementation of the PRECISION program at the site (e.g., Did AIRQ help you identify patients who were at risk for adverse health outcomes from their asthma that you would have otherwise missed?)
Time Frame: as for outcome 1
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Sites
  Yes | 5 | 3 | 1 | 9
  No | 1 | 3 | 0 | 4

4. Primary Outcome: Percentage Endorsement of Responses by Site HCPs for Each Categorical Item on the Post-study Survey Relating to Most and Least Helpful Parts of AIRQ
Description: The post-study HCP survey includes questions regarding the implementation of the PRECISION program at the site (e.g., What did you find most useful about AIRQ?)
Time Frame: as for outcome 1
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Sites
  What did you find most useful about AIRQ?: Total AIRQ® score | 4 | 1 | 1 | 6
  What did you find most useful about AIRQ?: Questions on impact/impairment (#1-6) | 2 | 0 | 0 | 2
  What did you find most useful about AIRQ?: Question on control (#7) | 0 | 0 | 0 | 0
  What did you find most useful about AIRQ?: Questions on exacerbations and healthcare resource utilization (#8-10) | 0 | 5 | 0 | 5
  What did you find least useful about AIRQ?: Total AIRQ® score | 0 | 0 | 0 | 0
  What did you find least useful about AIRQ?: Questions on impact/impairment (#1-6) | 0 | 4 | 0 | 4
  What did you find least useful about AIRQ?: Question on control (#7) | 2 | 2 | 0 | 4
  What did you find least useful about AIRQ?: Questions on exacerbations and healthcare resource utilization (#8-10) | 4 | 0 | 1 | 5

5. Primary Outcome: Percentage Endorsement of Responses by Site HCPs for the Categorical Item on the Post-study Survey Relating to Frequency of Referring to a Specialist or Practice Type Different Than Their Own While Using the AIRQ
Description: The post-study HCP survey includes questions regarding the implementation of the PRECISION program at the site (e.g., While using AIRQ how often did you refer to a specialist or practice type different than your own?)
Time Frame: as for outcome 1
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Sites
  No different than if I did not have the tools | 2 | 6 | 1 | 9
  More often than before | 4 | 0 | 0 | 4
  Less often than before | 0 | 0 | 0 | 0

6. Primary Outcome: Percentage Endorsement of Responses by Site HCPs for the Categorical Item on the Post-study Survey Relating to Components of Care Improved by AIRQ
Description: The post-study HCP survey includes questions regarding the implementation of the PRECISION program at the site (e.g., Did AIRQ improve any of the following?)
Time Frame: as for outcome 1
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Sites
  Increased recognition of patients whose asthma placed their health at risk | 4 | 4 | 1 | 9
  Increased recognition of conditions/risks, comorbidities driving poor asthma control | 5 | 1 | 0 | 6
  Improved recognition of patient goals | 3 | 3 | 1 | 7
  Improved patient engagement with their treatment, risk, or control | 5 | 4 | 1 | 10
  Improved efficiency of patient telehealth visit | 2 | 2 | 0 | 4
  Improved efficiency of in-person asthma clinic visit | 2 | 1 | 0 | 3
  Increased educational efforts | 6 | 3 | 1 | 10

7. Primary Outcome: Percentage Endorsement of Responses by Site HCPs for Each Categorical Item on the Post-study Survey Relating to Importance of Using Different Components of the PRECISION Program
Description: The post-study HCP survey includes questions regarding the implementation of the PRECISION program at the site (e.g., How important was it for you to use the Assess component of the Asthma Checklist (page 1) with the AIRQ?).
Time Frame: as for outcome 1
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Sites
  How important was it for you to use the Assess component of the Asthma Checklist with the AIRQ?: Very important | 4 | 0 | 0 | 4
  How important was it for you to use the Assess component of the Asthma Checklist with the AIRQ?: Somewhat important | 2 | 5 | 1 | 8
  How important was it for you to use the Assess component of the Asthma Checklist with the AIRQ?: Not at all important | 0 | 1 | 0 | 1
  How important was it for you to use the Assess component of the Asthma Checklist with the AIRQ?: Did not use | 0 | 0 | 0 | 0
  How important was it for you to use the Adjust and Review components of the Asthma Checklist?: Very important | 3 | 0 | 0 | 3
  How important was it for you to use the Adjust and Review components of the Asthma Checklist?: Somewhat important | 2 | 5 | 1 | 8
  How important was it for you to use the Adjust and Review components of the Asthma Checklist?: Not at all important | 0 | 0 | 0 | 0
  How important was it for you to use the Adjust and Review components of the Asthma Checklist?: Did not use | 1 | 1 | 0 | 2
  How important would it be for PCPs to use the Asthma Checklist Assess component with the AIRQ?: Very important | 5 | 3 | 1 | 9
  How important would it be for PCPs to use the Asthma Checklist Assess component with the AIRQ?: Somewhat important | 1 | 3 | 0 | 4
  How important would it be for PCPs to use the Asthma Checklist Assess component with the AIRQ?: Not at all important | 0 | 0 | 0 | 0
  How important would it be for PCPs to use the Asthma Checklist Assess component with the AIRQ?: Did not use | 0 | 0 | 0 | 0
  How important would it be for Specialists to use Asthma Checklist Adjust/Review pages with AIRQ?: Very important | 2 | 1 | 0 | 3
  How important would it be for Specialists to use Asthma Checklist Adjust/Review pages with AIRQ?: Somewhat important | 3 | 4 | 1 | 8
  How important would it be for Specialists to use Asthma Checklist Adjust/Review pages with AIRQ?: Not at all important | 0 | 1 | 0 | 1
  How important would it be for Specialists to use Asthma Checklist Adjust/Review pages with AIRQ?: Did not use | 1 | 0 | 0 | 1
  How important would it be for Non-prescribers to use Asthma Checklist Assess component with AIRQ?: Very important | 3 | 3 | 0 | 6
  How important would it be for Non-prescribers to use Asthma Checklist Assess component with AIRQ?: Somewhat important | 3 | 3 | 1 | 7
  How important would it be for Non-prescribers to use Asthma Checklist Assess component with AIRQ?: Not at all important | 0 | 0 | 0 | 0
  How important would it be for Non-prescribers to use Asthma Checklist Assess component with AIRQ?: Did not use | 0 | 0 | 0 | 0

8. Primary Outcome: Average Number of Patients Treated Using the PRECISION Program at Each Site as Reported by Site HCPs by Site Type
Description: The post-study HCP survey asks sites to report the number of patients treated using the PRECISION program at their site. One HCP per site reported on the number of patients treated using the PRECISION program at their site. The mean presented is the number of patients at each site as reported by site HCPs divided by the number of sites.
Time Frame: as for outcome 1
Population: Number of site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Mean (Standard Deviation); unit: Patients per site
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites | Specialty Care Sites | Novelty Care Site | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Number analyzed (Sites) | 6 | 6 | 1 | 13
Patients per site | 72.2 (25.9) | 46.2 (35.5) | 130.0 (NA) — There is no standard deviation because there is only 1 site | 64.6 (36.9)

9. Primary Outcome: Descriptive Free-text Site HCP Responses to Open-ended Question on Post-study Survey on Features of PRECISION Program: Primary Care Sites
Description: On the post-study survey, one HCP per site (site PI) was asked to describe the features of the PRECISION program they thought were the most useful and could be improved when implemented at their site
Time Frame: Post-study survey was completed between 32.9 weeks and 50.6 weeks of last patient end of follow-up across sites; end of follow up was 36 weeks from last patient enrolled at site.
Population: Number of primary care site HCPs who responded to the post-study HCP survey (one HCP responded for each site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites
Number analyzed (Participants) | 6
Number analyzed (Sites) | 6
Sites
  Most useful features: Helped bring asthma and asthma control to the forefront | 2
  Most useful features: Closer attention paid to use of inhalers | 2
  Most useful features: Improved asthma patient care | 2
  Most useful features: Provided objective numerical score to discuss with patients | 1
  Most useful features: Helped patients understand their asthma status | 1
  Features to be improved: Patient self-completing AIRQ prior to visit, possibly as self-assessment | 2
  Features to be improved: AIRQ mode of incorporation into workflow | 2
  Features to be improved: Stylistic features of AIRQ and Asthma checklist | 2
  Features to be improved: Assess patients not on optimal inhalers due to medication unaffordability | 1

10. Primary Outcome: Descriptive Free-text Site HCP Responses to Open-ended Question on Post-study Survey on Features of PRECISION Program: Specialty Care Sites
Description: On the post-study survey, one HCP per site (site PI) was asked to describe the features of the PRECISION program they thought were most useful and could be improved when implemented at their site
Time Frame: Post-study survey was completed between 22.1 weeks and 50.4 weeks of last patient end of follow-up across sites; end of follow up was 36 weeks from last patient enrolled at site.
Population: Number of speciality care site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Specialty Care Sites
Number analyzed (Participants) | 6
Number analyzed (Sites) | 6
Sites
  Most useful features: Improved recognition of asthma control and risk | 3
  Most useful features: Ease of administration of AIRQ | 2
  Most useful features: Improved recognition of how patients assess their asthma | 1
  Most useful features: Patient educational goals | 1
  Features to be improved: Ease of implementation in workflow | 3
  Features to be improved: More detailed questions on AIRQ | 1
  Features to be improved: Redundancy of Asthma Checklist | 1

11. Primary Outcome: Descriptive Free-text Site HCP Responses to Open-ended Question on Post-study Survey on Features of PRECISION Program: Novel Care Site
Description: as for outcome 10
Time Frame: Post-study survey was completed 5 weeks after last patient end of follow-up; end of follow up was 6 weeks from last patient enrolled at site.
Population: Number of novel care site HCPs who responded to the post-study HCP survey (one HCP responded per site)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Groups:
- Novel Care Site: e.g., telehealth component of Allergy and Asthma Network
Arm/Group | Novel Care Site
Number analyzed (Participants) | 1
Number analyzed (Sites) | 1
Sites
  Most useful features: Educational resources | 1
  Features to be improved: Adding additional response options for the AIRQ rescue inhaler use question | 1

12. Primary Outcome: Descriptive Free-text Clinician Responses to the Qualitative Interview Questions on Implementation and Features of the Asthma Precision Program: Primary Care Sites
Description: Site clinicians were asked to respond to several open-ended questions regarding background information about the site, the implementation process at their site, use of the Asthma Checklist and educational resources, and feedback on the entire program.
Time Frame: Post-study clinician interviews were completed between -2 weeks (interviews completed a little sooner than end of follow-up) and 52.4 weeks of last patient end of follow-up across sites; end of follow up was 36 weeks from last patient enrolled at site.
Population: Number of clinicians from primary care sites who took part in the interviews (more than one clinician per site took part in the interviews)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites
Number analyzed (Participants) | 7
Number analyzed (Sites) | 6
Sites
  Benefits: Helped with assessing asthma control and risk | 4
  Benefits: Helped optimize care | 3
  Benefits: Helped guide treatment decisions | 3
  Benefits: Helped improve patient assessment and self-management | 4
  Benefits: Providing educational resources was valuable for patient and staff education | 3
  Benefits: AIRQ preferred over other screening tools | 1
  Benefits: AIRQ score confirmed and reassured patient of need for referral | 1
  Benefits: Increased provider and patient accountability for Asthma prevention | 1
  Ease of implementation: Easy to use | 5
  Ease of implementation: AIRQ questionnaire was quick to complete | 1
  Ease of implementation: Patients needing assistance to complete the AIRQ questions | 1
  Ease of implementation: Difficulty accessing and using the website | 2
  Ease of implementation: Additional demands to implement the AIRQ | 1
  Barriers to implementation: Busy HCP schedules | 6
  Barriers to implementation: Difficulty sharing AIRQ questionnaire in Telehealth visits | 3
  Barriers to implementation: COVID-related challenges | 2
  Barriers to implementation: Interest in several medical conditions, not just Asthma | 1
  Areas for improvement: Ease process of incorporating AIRQ into workflow | 3
  Areas for improvement: Facilitate patient access and completion of the AIRQ prior to the visit | 3
  Areas for improvement: Incorporate into EMR | 4
  Areas for improvement: Support with printing the AIRQ forms in color | 2
  Areas for improvement: Improve website to make it more user friendly | 1
  Areas for improvement: Translate AIRQ into other languages | 1
  Areas for improvement: Allow insurance coverage for time spent administering AIRQ | 1

13. Primary Outcome: Descriptive Free-text Key Site Staff Responses to the Qualitative Interview Questions on Implementation and Features of the Asthma Precision Program: Primary Care Sites
Description: Key site staff were asked to respond to several open-ended questions regarding background information about the site, the implementation process at their site, use of the Asthma Checklist and educational resources, and feedback on the entire program.
Time Frame: Post-study key site staff interviews were completed between -2 weeks (interviews completed a little sooner than end of follow-up) and 43 weeks of last patient end of follow-up across sites; end of follow up was 36 weeks from last patient enrolled at site.
Population: Number of key site staff from primary care sites who took part in the interviews (one key site staff per site took part in the interviews)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites
Number analyzed (Participants) | 5
Number analyzed (Sites) | 5
Sites
  Benefits: Opened up discussion with patients to improve Asthma care | 2
  Benefits: Brought Asthma to the forefront | 2
  Benefits: Improved detection of Asthma problems | 1
  Benefits: Doing more Asthma action plans | 1
  Benefits: Making greater use of pharmacy students to educate and support patients | 1
  Ease of implementation: Time added to workflow | 4
  Ease of implementation: AIRQ questionnaire straightforward to complete | 3
  Ease of implementation: AIRQ questionnaire quick to complete | 2
  Ease of implementation: Asthma Checklist difficult to use | 2
  Ease of implementation: Need to review AIRQ answers with patients due to incorrect answers | 1
  Ease of implementation: Additional demands to implement the AIRQ | 1
  Ease of implementation: Need for supplemental readily accessible materials | 1
  Ease of implementation: Factors that eased implementation | 1
  Barriers to implementation: Rescheduled or cancelled appointments | 3
  Barriers to implementation: Busy HCP schedules | 2
  Barriers to implementation: AIRQ not presented as part of regular medical visit/workflow | 1
  Barriers to implementation: Asthma often trumped by other health concerns | 1
  Barriers to implementation: Issues with Asthma patient list | 1
  Barriers to implementation: Recommended procedures not always completed in telehealth visits | 1
  Barriers to implementation: More difficult to do hands-on teaching in telehealth visits | 1
  Areas for improvement: Incorporating AIRQ as part of regular medical visit | 1
  Areas for improvement: Incorporating AIRQ in EMR | 1
  Areas for improvement: Having an electronic fillable version of the AIRQ | 1
  Areas for improvement: Recall period for AIRQ | 1
  Areas for improvement: Removing unnecessary questions on AIRQ | 1
  Areas for improvement: Restructuring the checklist | 1

14. Primary Outcome: Descriptive Free-text Clinician Responses to the Qualitative Interview Questions on Implementation and Features of the Asthma Precision Program: Specialty Care Sites
Description: Site clinicians were asked to respond to several open-ended interview questions regarding background information about the site, the implementation process at their site, use of the Asthma Checklist and educational resources, and feedback on the entire program.
Time Frame: Post-study clinician interviews were completed between -6.3 weeks (interviews completed a little sooner than end of follow-up) and 23 weeks of last patient end of follow-up across sites; end of follow up was 36 weeks from last patient enrolled at site.
Population: Number of clinicians from specialty care sites who took part in the interviews (more than one clinician per site took part in the interviews)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Specialty Care Sites
Number analyzed (Participants) | 7
Number analyzed (Sites) | 6
Sites
  Benefits: Helped with assessing asthma control and risk | 6
  Benefits: AIRQ preferred by HCP over other screening tools | 4
  Benefits: Helped optimize care | 3
  Benefits: AIRQ questionnaire guided treatment recommendations | 2
  Benefits: AIRQ questionnaire helped improve patient assessment and self-management | 2
  Benefits: Comprehensive Asthma management tool | 1
  Benefits: AIRQ questionnaire could be used to check on whether a full medical visit is needed | 1
  Benefits: Aligns with clinician's approach of assessing Asthma | 1
  Ease of implementation: Easy to use | 5
  Ease of implementation: Difficulty accessing and using the website | 3
  Ease of implementation: AIRQ educational materials too complex for the patient's education level | 1
  Barriers to implementation: Busy HCP schedules | 3
  Barriers to implementation: Difficulty administering AIRQ questionnaire in Telehealth visits | 2
  Barriers to implementation: Not sharing educational resources to not overburden patients | 1
  Barriers to implementation: Cannot find a way to implement automated distribution of AIRQ | 1
  Barriers to implementation: Difficulty combining additional with existing resources | 1
  Barriers to implementation: ACT required by insurance companies to renew biologics; hard to do both | 1
  Areas for improvement: Making Asthma Checklist and educational resources more easily accessible | 1
  Areas for improvement: Incorporating into the EMR | 1
  Areas for improvement: Supporting automated distribution of AIRQ | 1
  Areas for improvement: Building AIRQ into an app for automatic notification of Asthma complications | 1
  Areas for improvement: Making the educational materials available on an app as opposed to website | 1
  Areas for improvement: Making the educational materials easier to understand | 1
  Areas for improvement: Would be useful to share the tools with other HCPs | 1

15. Primary Outcome: Descriptive Free-text Key Site Staff Responses to the Qualitative Interview Questions on Implementation and Features of the Asthma Precision Program: Specialty Care Sites
Description: as for outcome 13
Time Frame: Post-study site staff interviews were completed between -6.3 weeks (interviews completed a little sooner than end of follow-up) and 4.7 weeks of last patient end of follow-up across sites; end of follow up was 36 weeks from last patient enrolled at site.
Population: Number of key site staff from specialty care sites who took part in the interviews (one key site staff per site took part in the interviews)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Specialty Care Sites
Number analyzed (Participants) | 2
Number analyzed (Sites) | 2
Sites
  Benefits: Great tool to evaluate patients | 1
  Ease of implementation: Time consuming process | 1
  Ease of implementation: AIRQ questionnaire quick to complete | 1
  Ease of implementation: Needing to ensure patients respond correctly to the AIRQ | 1
  Barriers to implementation: Ensuring clinicians' schedule was not interrupted when implementing AIRQ | 1
  Barriers to implementation: Difficulty transmitting AIRQ results between HCP, patient, site staff | 1
  Areas for improvement: Recall period for AIRQ | 1

16. Primary Outcome: Descriptive Free-text HCP Responses to the Qualitative Interview Questions on Implementation and Features of the Asthma Precision Program: Novel Site
Description: Site HCPs were asked to respond to several open-ended interview questions regarding background information about the site, the implementation process at their site, use of the Asthma Checklist and educational resources, and feedback on the entire program.
Time Frame: Post-study HCP interviews were completed 5 weeks after last patient end of follow-up; end of follow up was 6 weeks from last patient enrolled at site.
Population: Number of HCPs from novel site who took part in the interviews
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Novel Site
Number analyzed (Participants) | 1
Number analyzed (Sites) | 1
Sites
  Benefits: AIRQ tools helped with assessing asthma control and risk | 1
  Benefits: Preferred over other screening tools | 1
  Benefits: Helped optimize care | 1
  Benefits: Providing educational resources post visit was valuable for patient and staff education | 1
  Benefits: Resources were empowering for patients | 1
  Ease of implementation: Easy to use | 1
  Ease of implementation: Quick to complete | 1
  Ease of implementation: Use of infographics | 1
  Ease of implementation: Difficulty using and accessing the website | 1
  Ease of implementation: Difficulty accessing and using the website | 1
  Barriers to implementation: None discussed | 0
  Areas for improvement: Revising question on use of rescue inhaler or nebulizer | 1

17. Primary Outcome: Descriptive Free-text Key Site Staff Responses to the Qualitative Interview Questions on Implementation and Features of the Asthma Precision Program: Novel Site
Description: as for outcome 13
Time Frame: Post-study key site staff interviews were completed 5 weeks after last patient end of follow-up; end of follow up was 6 weeks from last patient enrolled at site.
Population: Number of key site staff from novel site who took part in the interviews
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Novelty Care Site
Number analyzed (Participants) | 1
Number analyzed (Sites) | 1
Sites
  Benefits: Great tool to evaluate patients | 1
  Benefits: Providing educational resources was valuable for patient education | 1
  Ease of implementation: Easy to implement in Telehealth visits with other programs | 1

18. Primary Outcome: Descriptive Free-text Site Staff Responses to the Implementation Touchpoint Questions: Primary Care Sites (Month 1)
Description: At each touchpoint, site staff were asked to respond to questions about the implementation of the PRECISION program (e.g., what aspects of the study implementation are going well for your site?)
Time Frame: Month 1 after start of implementation
Population: Number of primary care key site staff who took part in the touchpoints at month 1 (one key site staff per site participated)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites
Number analyzed (Participants) | 2
Number analyzed (Sites) | 2
Sites
  Benefits: Improved management of asthma and treatment plan | 2
  Benefits: Improved ability to discuss asthma history with patients | 1
  Benefits: Improved documentation of patients' asthma, including triggers and exacerbations | 1
  Benefits: Helped assess asthma control and risk | 2
  Benefits: Patients are getting more asthma education through the use of the online resources | 1
  Ease of implementation: AIRQ questionnaire easily understood by patients | 1
  Ease of implementation: Challenges accessing website for resources | 1
  Barriers to implementation: Patients scheduled with doctors in study rather than preferred doctor | 1
  Barriers to implementation: Staffing issues affecting recruitment into the study | 1
  Areas of improvement: Adding more pictures to website resources and making them more interactive | 1
  Areas of improvement: AIRQ wording modified to ensure participants report Asthma-related issues | 1
  Other: Less actual asthma during study period with COVID masks | 1

19. Primary Outcome: Descriptive Free-text Site Staff Responses to the Implementation Touchpoint Questions: Primary Care Sites (Month 2)
Description: as for outcome 18
Time Frame: Month 2 after start of implementation
Population: Number of primary care key site staff who took part in the touchpoints at month 2 (one key site staff per site participated)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Primary Care Sites
Number analyzed (Participants) | 2
Number analyzed (Sites) | 2
Sites
  Benefits: Asthma Checklist allows for a more comprehensive discussion of patient's Asthma | 1
  Barriers to implementation: No challenges, just working with clinicians to set up study | 1
  Ease of implementation: Discrepancies between AIRQ exacerbation answers and medical chart | 1
  Ease of implementation: Wanting to integrate the website more to improve use | 1
  Ease of implementation: Need to simplify and standardize the execution of the AIRQ | 1
  Other: Looking into conducting more telehealth visits | 1
  Other: Opening it up to more providers | 1

20. Primary Outcome: Descriptive Free-text Site Staff Responses to the Implementation Touchpoint Questions: Specialty Care Sites (Month 1)
Description: as for outcome 18
Time Frame: Month 1 after start of implementation
Population: Number of specialty care key site staff who took part in the touchpoints at month 1 (one key site staff per site participated)
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Specialty Care Sites
Number analyzed (Participants) | 2
Number analyzed (Sites) | 2
Sites
  Benefits: AIRQ preferred over ACT by providers; gives additional information | 2
  Benefits: Helps follow-up on the low/med/high dose for the inhaled corticosteroids | 1
  Benefits: HCPs are engaged and like being involved in patient care | 1
  Benefits: Patients prefer the AIRQ scale over the ACT 5-point scale (like Yes/No items) | 1
  Ease of implementation: Patients (including adolescents) can easily complete the AIRQ on their own | 1
  Ease of implementation: Lead nurse training an additional site coordinator | 1
  Barriers to implementation: Website not found to be helpful in specialty care | 2
  Barriers to implementation: Issues with Sharepoint | 1
  Barriers to implementation: Staffing issues affecting recruitment and administration of AIRQ | 1

21. Primary Outcome: Descriptive Free-text Site Staff Responses to the Implementation Touchpoint Questions: Novel Care Site (Month 2)
Description: as for outcome 18
Time Frame: Month 2 after start of implementation
Population: Number of novelty care key site staff who took part in the touchpoints at month 2
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Novelty Care Site
Number analyzed (Participants) | 1
Number analyzed (Sites) | 1
Sites
  Benefits: None discussed | 0
  Ease of implementation: AIRQ is easy to implement and very self-explanatory | 1
  Ease of implementation: Graphics of educational materials are helpful for HCPs and patients | 1
  Barriers to implementation: Recruitment slower than expected; patients moving away from telehealth | 1
  Barriers to implementation: Difficult to collect exacerbation history; no access to patient files | 1
  Areas for improvement: Sending participants the AIRQ ahead of the call to ease administration | 1

22. Secondary Outcome: Change in Patient AIRQ Score From Baseline to Follow-up Visits: Mean and Standard Deviation at Each Visit
Description: AIRQ scores range from 0 to 10, where lower scores indicate more well-controlled asthma
  The AIRQ was used for the initial study visit, and a follow-up AIRQ that employs the same 10 questions as the AIRQ but for the 3 risk questions where exacerbation history covers a 3 month look-back period instead of a 12 month look-back period was used for follow-up visits.
Time Frame: Mean (SD) time to follow-up was 3.3 (SD = 1.4) months
Population: Number of patients with a baseline and follow-up visit
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Primary Care: e.g., private practice, FQHC
- Specialty Care: e.g., pulmonary, asthma/immunology
Arm/Group | Primary Care | Specialty Care | Novel Site
Number analyzed (Participants) | 145 | 100 | 126
Points
  Baseline AIRQ Score | 1.8 (2.15) | 4.2 (3.15) | 4.5 (2.89)
  Follow-up AIRQ Score | 1.1 (1.84) | 3.1 (3.35) | 2.8 (2.56)

23. Secondary Outcome: Change in Patient AIRQ Score From Baseline to Follow-up Visits: Mean Difference and Confidence Interval
Description: as for outcome 22
Time Frame: Mean (SD) time to follow-up was 3.3 (SD = 1.4) months
Population: Number of patients with a baseline and follow-up visit
Measure: Mean (95% Confidence Interval); unit: Points
Arm/Group | Primary Care | Specialty Care | Novel Site
Number analyzed (Participants) | 145 | 100 | 126
Points | -0.7 [-1.00 to -0.40] | -1.1 [-1.55 to -0.67] | -1.7 [-2.20 to -1.28]

24. Secondary Outcome: Change in Patient AIRQ Control Level From Baseline to Follow-up Visit
Description: AIRQ Control level can be categorized as "well controlled", "not-well controlled" or "very poorly controlled"
  The AIRQ was used for the initial study visit, and a follow-up AIRQ that employs the same 10 questions as the AIRQ but for the 3 risk questions where exacerbation history covers a 3 month look-back period instead of a 12 month look-back period was used for follow-up visits.
Time Frame: Mean (SD) time to follow-up was 3.3 (SD = 1.4) months
Population: Number of patients in each AIRQ control level category at follow-up by AIRQ control level category at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care | Specialty Care | Novel Site
Number analyzed (Participants) | 145 | 100 | 126
Participants
  Baseline AIRQ control category: Well controlled: number analyzed (Participants) | 81 | 24 | 23
  Baseline AIRQ control category: Well controlled: Follow-up AIRQ Control Category: Well controlled (0-1) | 75 | 23 | 20
  Baseline AIRQ control category: Well controlled: Follow-up AIRQ Control Category: Not well controlled (2-4) | 4 | 0 | 2
  Baseline AIRQ control category: Well controlled: Follow-up AIRQ Control Category: Very poorly controlled (5-10) | 2 | 1 | 1
  Baseline AIRQ control category: Not well controlled: number analyzed (Participants) | 45 | 36 | 39
  Baseline AIRQ control category: Not well controlled: Follow-up AIRQ Control Category: Well controlled (0-1) | 23 | 23 | 17
  Baseline AIRQ control category: Not well controlled: Follow-up AIRQ Control Category: Not well controlled (2-4) | 18 | 9 | 16
  Baseline AIRQ control category: Not well controlled: Follow-up AIRQ Control Category: Very poorly controlled (5-10) | 4 | 4 | 6
  Baseline AIRQ control category: Very poorly controlled: number analyzed (Participants) | 19 | 40 | 64
  Baseline AIRQ control category: Very poorly controlled: Follow-up AIRQ Control Category: Well controlled (0-1) | 6 | 5 | 15
  Baseline AIRQ control category: Very poorly controlled: Follow-up AIRQ Control Category: Not well controlled (2-4) | 6 | 6 | 24
  Baseline AIRQ control category: Very poorly controlled: Follow-up AIRQ Control Category: Very poorly controlled (5-10) | 7 | 29 | 25

25. Secondary Outcome: Percentage of Endorsement of Responses for Each of the 8 Categorical Items on the ACE Questionnaire
Description: The ACE questionnaire includes 8 items each with Likert scale responses (strongly agree, agree, disagree, strongly disagree). Participants completed this measure via a patient web survey.
Time Frame: Baseline
Population: Number of patients who completed the patient web-survey which was optional to patients who took part in the study
Measure: Count of Participants; unit: Participants
Groups:
- Novelty Care: e.g., telehealth component of Allergy and Asthma Network
Arm/Group | Primary Care | Specialty Care | Novelty Care
Number analyzed (Participants) | 67 | 31 | 9
Participants
  Item 1 (The AIRQ helped me discuss my asthma with my health care provider(s).): Strongly Agree | 26 | 7 | 6
  Item 1 (The AIRQ helped me discuss my asthma with my health care provider(s).): Agree | 29 | 17 | 2
  Item 1 (The AIRQ helped me discuss my asthma with my health care provider(s).): Disagree | 6 | 4 | 1
  Item 1 (The AIRQ helped me discuss my asthma with my health care provider(s).): Strongly Disagree | 0 | 1 | 0
  Item 1 (The AIRQ helped me discuss my asthma with my health care provider(s).): Not applicable | 1 | 0 | 0
  Item 1 (The AIRQ helped me discuss my asthma with my health care provider(s).): Missing | 5 | 2 | 0
  Item 2 (I received information about my asthma that helped me better understand my condition.): Strongly Agree | 24 | 10 | 5
  Item 2 (I received information about my asthma that helped me better understand my condition.): Agree | 27 | 17 | 3
  Item 2 (I received information about my asthma that helped me better understand my condition.): Disagree | 8 | 2 | 1
  Item 2 (I received information about my asthma that helped me better understand my condition.): Strongly Disagree | 2 | 0 | 0
  Item 2 (I received information about my asthma that helped me better understand my condition.): Not applicable | 1 | 0 | 0
  Item 2 (I received information about my asthma that helped me better understand my condition.): Missing | 5 | 2 | 0
  Item 3 (I received information about my asthma medications.): Strongly Agree | 21 | 10 | 6
  Item 3 (I received information about my asthma medications.): Agree | 23 | 15 | 1
  Item 3 (I received information about my asthma medications.): Disagree | 16 | 4 | 1
  Item 3 (I received information about my asthma medications.): Strongly Disagree | 1 | 0 | 0
  Item 3 (I received information about my asthma medications.): Not applicable | 0 | 0 | 1
  Item 3 (I received information about my asthma medications.): Missing | 6 | 2 | 0
  Item 4 (My health care providers explained the results of tests that I have taken for my asthma.): Strongly Agree | 20 | 12 | 4
  Item 4 (My health care providers explained the results of tests that I have taken for my asthma.): Agree | 16 | 12 | 1
  Item 4 (My health care providers explained the results of tests that I have taken for my asthma.): Disagree | 3 | 0 | 2
  Item 4 (My health care providers explained the results of tests that I have taken for my asthma.): Strongly Disagree | 0 | 0 | 1
  Item 4 (My health care providers explained the results of tests that I have taken for my asthma.): Not applicable | 23 | 5 | 1
  Item 4 (My health care providers explained the results of tests that I have taken for my asthma.): Missing | 5 | 2 | 0
  Item 5 (I was told the reason why tests for my asthma were ordered.): Strongly Agree | 26 | 13 | 5
  Item 5 (I was told the reason why tests for my asthma were ordered.): Agree | 15 | 9 | 0
  Item 5 (I was told the reason why tests for my asthma were ordered.): Disagree | 3 | 1 | 2
  Item 5 (I was told the reason why tests for my asthma were ordered.): Strongly Disagree | 1 | 0 | 0
  Item 5 (I was told the reason why tests for my asthma were ordered.): Not applicable | 17 | 6 | 2
  Item 5 (I was told the reason why tests for my asthma were ordered.): Missing | 5 | 2 | 0
  Item 6 (I was given information about additional care that I need for my asthma.): Strongly Agree | 21 | 12 | 5
  Item 6 (I was given information about additional care that I need for my asthma.): Agree | 23 | 9 | 0
  Item 6 (I was given information about additional care that I need for my asthma.): Disagree | 5 | 2 | 2
  Item 6 (I was given information about additional care that I need for my asthma.): Strongly Disagree | 0 | 0 | 0
  Item 6 (I was given information about additional care that I need for my asthma.): Not applicable | 13 | 6 | 2
  Item 6 (I was given information about additional care that I need for my asthma.): Missing | 5 | 2 | 0
  Item 7 (I was included in making decisions about my asthma treatment.): Strongly Agree | 38 | 18 | 5
  Item 7 (I was included in making decisions about my asthma treatment.): Agree | 20 | 11 | 2
  Item 7 (I was included in making decisions about my asthma treatment.): Disagree | 4 | 0 | 0
  Item 7 (I was included in making decisions about my asthma treatment.): Strongly Disagree | 0 | 0 | 1
  Item 7 (I was included in making decisions about my asthma treatment.): Not applicable | 0 | 0 | 1
  Item 7 (I was included in making decisions about my asthma treatment.): Missing | 5 | 2 | 0
  Item 8 (Time spent with health care provider(s) today discussing my asthma was better.): Strongly Agree | 22 | 9 | 4
  Item 8 (Time spent with health care provider(s) today discussing my asthma was better.): Agree | 34 | 11 | 3
  Item 8 (Time spent with health care provider(s) today discussing my asthma was better.): Disagree | 6 | 8 | 1
  Item 8 (Time spent with health care provider(s) today discussing my asthma was better.): Strongly Disagree | 0 | 0 | 0
  Item 8 (Time spent with health care provider(s) today discussing my asthma was better.): Not applicable | 0 | 0 | 0
  Item 8 (Time spent with health care provider(s) today discussing my asthma was better.): Missing | 5 | 3 | 1

ADVERSE EVENTS:
Description: Adverse events were not collected as part of this study
Groups:
- Novel Care Sites: e.g., telehealth component of Allergy and Asthma Network
Arm/Group | Primary Care Sites | Specialty Care Sites | Novel Care Sites
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to low participation on the optional patient web-survey, limited data were available for the ACE, thus limiting full analyses of the secondary objective relating to patient satisfaction with visit when AIRQ implemented based on responses to ACE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Receiving party will keep Confidential Information in confidence and will not, at any time during or for ten years after the expiration of this Agreement, without the disclosing party's prior written consent, disclose, publish, disseminate or otherwise make available, any item of Confidential Information to any third party. Receiving party will use the Confidential Information only in connection with performance or receipt of Services, or in the exercise of a right granted under this Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT04891978/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT04891978/SAP_001.pdf